CLINICAL TRIAL: NCT00106795
Title: Assessing the Relationship Between Fatigue and Mitochondrial Toxicity in Patients With HIV/AIDS
Brief Title: Relationship Between Fatigue and Mitochondrial Damage in Patients With HIV/AIDS
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050127; 05-I-0127
Record Dates: First submitted 2005-03-30; First posted 2005-03-31 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2014-04-10

CONDITIONS: HIV Infections; Fatigue; HIV Positive; AIDS; Healthy Volunteer; HV
Keywords: Antiretrovirals; Adipocytes; Skeletal Muscle; Fatigue; HIV; AIDS; Lymphocytes; Lipodystrophy; HIV Positive; Healthy Volunteer; HV
MeSH Terms: conditions — HIV Infections; Fatigue; HIV Seropositivity; Acquired Immunodeficiency Syndrome; Lipodystrophy

SUMMARY:
This study will examine abnormalities in mitochondria (energy-producing machinery of cells) and in genes related to mitochondria in the blood cells, muscle, and fat of HIV-positive patients who are taking nucleoside reverse transcriptase inhibitors (NRTIs) and in patients not currently taking HIV medications, and compare the results to healthy volunteers. Many patients with HIV infection take NRTIs to help control the infection. These medications may damage cell mitochondria, possibly causing side effects such as fatigue. This study will explore the relationship between changes in mitochondria and related genes and patient reports of energy level, mood and quality of life.

Healthy volunteers and HIV-infected patients between 18 and 55 years of age may be eligible for this study. Healthy volunteers must test negative for the HIV antibody. HIV-positive patients must have been diagnosed positive for at least 1 year. Patients who are taking antiretroviral therapy must have been taking the same drug regimen (with at least two NTRIs and no protease inhibitors) for at least 3 months. HIV positive patients not taking antiretroviral medication must not have had antiretroviral therapy for at least 1 year. Candidates are screened with a medical history, brief physical examination, blood and urine tests, and questionnaires related to mood and energy.

Qualified volunteers will undergo the following procedures during three or four study visits:

Visit 1

Complete history and physical examination, blood tests, and questionnaires about energy level, mood, and quality of life.

Visit 2

Muscle and fat biopsy: Before the biopsy, blood is drawn to check blood counts and to test for pregnancy in women who can become pregnant. The biopsy is done on an outpatient basis in the operating room. The site of the biopsy (an area on the upper arm or upper leg) is numbed with an injection under the skin. A 1-inch incision is made over the muscle to be biopsied and a small sample of muscle tissue and small sample of fat are removed. The incision is then closed and bandaged. Following the biopsy, you will be monitored for about 4 hours in the clinic. Strenuous physical activity should be restricted in the week following biopsy to allow healing.

Visit 3

Examination of biopsy site and possible apheresis: The biopsy site is examined for healing. Apheresis may be scheduled for this visit or for an extra visit between the biopsy and the final visit. This procedure for obtaining white blood cells for study is optional. For apheresis, blood is withdrawn from a needle placed in a vein in the arm and the white cells are separated from the rest of the blood. The white cells are extracted and the red cells and plasma are then returned to the body through a second needle.

DETAILED DESCRIPTION:
Both HIV infection and antiretroviral nucleoside analogues (nucleoside reverse transcriptase inhibitors or NRTIs) are known to affect mitochondrial DNA content and mitochondrial function. A number of important clinical syndromes observed in HIV-infected persons relate to mitochondrial dysfunction including lactic acidosis, myopathy, cardiomyopathy, pancreatitis, peripheral neuropathy, and possibly lipodystrophy. Fatigue, one of the most prevalent complaints among persons with HIV infection, may also be the result of mitochondrial toxicity, though this has not been clearly established.

Availability of minimally invasive tests to assess mitochondrial toxicity would greatly facilitate understanding of the contribution of mitochondrial dysfunction to clinical syndromes. Mitochondrial dysfunction ultimately results in lactic acidosis; however, venous lactate measurements are neither adequately sensitive nor specific for identification of early mitochondrial dysfunction. Muscle and liver biopsies are currently considered to be the reference standards for the evaluation and diagnosis of mitochondrial toxicity in muscle and liver, but these invasive tests are impractical for routine and repeated evaluations. The recent development of a real-time polymerase chain reaction (PCR) assay to accurately quantify the mtDNA copy numbers per cell in peripheral blood mononuclear cells (PBMCs) may allow non-invasive assessment of mitochondrial toxicity. This technique has been applied in a limited fashion to muscle, adipose tissue and liver samples as well.

This pilot study seeks to examine the relationship between fatigue and other clinical parameters and markers of mitochondrial dysfunction. The goals of this study are threefold: 1) to investigate the relationship between subjective fatigue ratings and mitochondrial dysfunction through measurements of mtDNA depletion in skeletal muscle 2) to determine whether there is a relationship between evidence of mitochondrial dysfunction in muscle and evidence of mitochondrial dysfunction in lymphocytes or adipose tissue suggesting that examination of lymphocytes or adipose tissue may be adequate for the accurate diagnosis of mitochondrial dysfunction and 3) to identify genes and proteins as potential biomarkers for fatigue and mitochondrial toxicity. For this cross-sectional study, three groups of participants will be enrolled: HIV positive patients on NRTI-containing and protease-inhibitor sparing regimens (n=30), HIV patients currently taking no antiretroviral medications (n=30) and healthy controls (n=15). HIV patients on NRTIs will be stratified according to their fatigue level (0-3, 4-7 or 8-10). Participants will complete a battery of questionnaires regarding fatigue and undergo muscle and adipose tissue biopsy.

ELIGIBILITY:
* INCLUSION CRITERIA:

Men and women, ages 18-55 years, will be considered as potential candidates for this study.

Persons older than 55 years of age are excluded because of age related declines in mitochondrial number that may confound study results.

Ability to understand and provide informed consent.

Willing and able to comply with study requirements and procedures including storage of blood, muscle and adipose tissue samples for use in future studies of HIV, AIDS, immune function, muscle or adipose tissue diseases or other related diseases.

No or currently controlled depression.

Negative serum pregnancy test for females at screening and within one week prior to muscle and adipose tissue biopsy.

Specific lab criteria:

* Absolute neutrophil count greater than 1000/mm(3).
* PT/INR less than or equal to 1.5, PTT less than 45 sec.
* Platelets greater than 75,000/mm(3).
* Hemoglobin greater than or equal to 10.0mg/dl.
* Serum creatinine less than or equal to 1.8mg/dl.
* AST and ALT less than 2 times the upper limit of normal.
* Thyroid stimulating hormone and free thyroxine within normal limits.
* Serum testosterone within normal limits or on adequate replacement.

Willing to avoid aspirin-containing medications or the non-steroidal anti-inflammatory drug piroxicam (Feldene) for 10 days prior to muscle and adipose tissue biopsy and willing to discontinue other nonsteroidal anti-inflammatory drugs 24 hours prior to biopsy.

For HIV negative volunteers:

Negative HIV-1 antibody testing

For HIV positive volunteers:

Established HIV diagnosis (documentation of HIV-1 infection by licensed ELISA testing and confirmed by Western Blot).

HIV infection present greater than or equal to 1 year.

For patients in the antiretroviral treated group, on a stable combination antiretroviral treatment regimen not containing a protease inhibitor for at least 3 months prior to protocol screening.

For patients in the non-ART group, no antiretroviral treatment for at least one year.

Under the care of a primary care physician.

EXCLUSION CRITERIA:

Unable to provide informed consent.

Unable to understand protocol required questionnaires including inability to comprehend English (the fatigue questionnaires have not been validated in languages other than English).

Pregnant or breast-feeding.

Current treatment with an ARV regimen containing a protease inhibitor.

Opportunistic infection requiring treatment.

Concurrent malignancy requiring cytotoxic chemotherapy or radiation therapy.

History of myopathy or myositis.

Untreated or uncontrolled depression by clinical history or as indicated by a score on the Beck's Depression Inventory of greater than or equal to 19.

Severe psychiatric disorder that would interfere with adherence to protocol requirements.

Severe sleep disturbance.

Current alcohol or substance abuse.

Diabetes mellitus requiring drug therapy.

Decompensated cardiac or pulmonary disease.

Current use or a history of treatment with interleukin-2, interferon-alpha or other investigational agent(s) within 6 months of protocol screening.

Corticosteroid, immunosuppressive or cytotoxic agent use within 90 days of trial screening.

Any medical condition for which the principal investigator feels muscle and adipose tissue biopsy may be contraindicated.

Allergy to lidocaine.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2005-03-22; Study Completion 2014-04-10

CONTACTS AND LOCATIONS:
Overall Officials: Caryn G Morse, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Brinkman K, ter Hofstede HJ, Burger DM, Smeitink JA, Koopmans PP. Adverse effects of reverse transcriptase inhibitors: mitochondrial toxicity as common pathway. AIDS. 1998 Oct 1;12(14):1735-44. doi: 10.1097/00002030-199814000-00004. No abstract available. PMID 9792373
- [Background] Lewis W, Dalakas MC. Mitochondrial toxicity of antiviral drugs. Nat Med. 1995 May;1(5):417-22. doi: 10.1038/nm0595-417. PMID 7585087
- [Background] John M, Moore CB, James IR, Nolan D, Upton RP, McKinnon EJ, Mallal SA. Chronic hyperlactatemia in HIV-infected patients taking antiretroviral therapy. AIDS. 2001 Apr 13;15(6):717-23. doi: 10.1097/00002030-200104130-00007. PMID 11371686